CLINICAL TRIAL: NCT00397592
Title: The Effect of Exogenous Growth Hormone on the Mobilization of Endothelial Progenitor Cells
Brief Title: Growth Hormone's Effect on Endothelial Progenitor Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 051212; 1515
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2007-07

CONDITIONS: Cardiovascular Disease
Keywords: Growth Hormone; Cardiovascular System; Endothelial Progenitor Cells
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Growth Hormone

SUMMARY:
To assess the effect of short-term low-dose growth hormone therapy on the mobilization of endothelial progenitor cells from the bone marrow within a group of healthy adults.

DETAILED DESCRIPTION:
We are proposing a pilot study to assess the effect of the administration of recombinant human growth hormone on the number of endothelial progenitor cells (EPC's) in the peripheral circulation. An increase in the number of EPC's is viewed as beneficial, as it has been postulated that they provide an endogenous repair mechanism to counteract endothelial injury. Additionally, a reduced number of EPC's has been found to independently predict atherosclerotic disease progression. Mechanisms proposed for enhancing the number of circulating EPC's and their function include an increase in proliferation, mobilization from the bone marrow, or prevention of EPC apoptosis. Thus, a pharmacologic manipulation of the number of EPC's in the peripheral circulation could potentially serve as a mechanism by which endothelial function, and thus vascular health, may be improved.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 thru 65
* Serum IGF-1 in the lower half of the age and gender-specific normal range at the time of screening visit

Exclusion Criteria:

* Systemic hypertension, as defined as current BP >140/90 on screening visit, or taking anti-hypertensive therapy.
* Diabetes mellitus, as defined by known diagnosis or Fasting Blood Glucose >126 at the time of screening visit.
* Women who are pregnant or nursing, as confirmed by history or seum beta-hCG at the time of screening visit.
* Women who are taking exogenous oral estrogens of any kind.
* Personal history of active cancer or recurrence within the past 10 years, with the exception of non-melanoma skin cancer.
* Personal history of an untreated benign intracranial neoplasm.
* Initiation of statin therapy during the course of the study.
* A serum IGF-1 level below the age and gender-specific normal range at the time of screening visit.
* Renal insufficiency, as defined by a GFR <60 mls/min/1.73 m2 upon Renal Function panel at the time of screening visit.
* Hepatic insufficiency, as defined by an AST and/or ALT >twice the upper limit of normal at the time of screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Number of Endothelial Progenitor Cells per mm^2 in culture after a maximum of 8 weeks of growth hormone therapy or until somatomedin-C is in the upper quartile of the normal range, as compared to baseline.

SECONDARY OUTCOMES:
All outcome measures will be assessed at baseline and following either a maximum of 8 weeks of growth hormone therapy or until somatomedin-C is in the upper quartile of the normal range:CD34/KDR+ Endothelial Progenitor Cells
Plasma nitrite and nitrate
L-Arginine
ADMA
estradiol
erythropoietin
SDF-1
VEGF

CONTACTS AND LOCATIONS:
Overall Officials: Doug Vaughan, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States